CLINICAL TRIAL: NCT06829810
Title: Long-term Outcomes of Glaucoma Surgery in a Real-life Setting: the Agora Registry Study
Acronym: GLAUCOSURG
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/89
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Intraocular pressure; glaucoma; ocular hypertension; glaucoma surgery; non penetrating deep sclerectomy; trabeculectomy; glaucoma drainage device
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Modelisation of intraocular pressure profile — Modelisation of IOP profile of all surgical techniques and additional procedures during the follow-up

SUMMARY:
Retrospective cohort study performed at Bordeaux University Hospital, which aims to analyze long-term safety and efficacy of different techniques of glaucoma surgery including filtering glaucoma surgeries, glaucoma drainage devices or minimally invasive glaucoma surgeries. All patients operated on in the department in the standard of care were proposed to be included in the AGORA registry study. The main outcome will be to define a modelisation of IOP profile based on the surgical technique. Secondary outcomes will be to analyze factors influencing IOP evolution as well as long-term safety and efficacy outcomes of the included surgical techniques.

DETAILED DESCRIPTION:
Glaucoma is a progressive degenerative optic neuropathy characterized by excavation of the optic nerve and the appearance, deepening and widening of visual field deficits (scotomas). It is the leading cause of irreversible blindness in France and worldwide. Although glaucoma is a progressive degenerative optic neuropathy with a multifactorial mechanism, all therapeutic studies have shown that lowering intraocular pressure (IOP) remains the only modulable causal factor that can stabilize or slow disease progression. It is also estimated that the glaucoma population requiring a surgery is approximately 5-10%. There is a wide range of surgical techniques for lowering IOP including filtering surgeries (trabeculectomy, non penetrating deep sclerectomy), glaucoma drainage devices and minimally invasive glaucoma surgeries. All these surgeries are acknowledged to reduce intraocular pressure but are also associated with risk of severe perioperative complications depending on glaucoma severity or ophthalmological characteristics. In addition some of them require additional procedures to maintain treatment success. These additional procedures are the consequence of IOP fluctuations over time following glaucoma surgeries. Although IOP is the main factors to control glaucoma over time, these real-life IOP fluctuations limit the use and the interpretability of survival analysis for long-term outcomes of each surgical procedure.

The aim of this study is to define a modelisation of IOP profile based on the surgical techniques and to analyze factors influencing IOP evolution as well as long-term safety and efficacy outcomes of the included surgical techniques. Demographical, ophthalmological, surgical parameters and all follow-up visits data will be collected in the standard of care of all patients who accepted to be included in the AGORA registry study. From November 2010 to April 2023, 2420 surgical procedures were recorded in the registry including 1584 Non penetrating deep sclerectomy, 212 trabeculectomy, 354 Istent or 95 high Intensity Focused Ultrasound. IOP evolution over time will be described for each surgical technique and a statistical model will be defined.

The modelisation of IOP with time and the description of risk factors of success or failure over the long-term of each surgical technique should help clinicians to make a more personalized surgical decision in order to maintain visual performances of glaucoma patients with time.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 with glaucoma or ocular hypertonia treated in the ophthalmology department of Bordeaux University Hospital between 2011 and 2022.

Exclusion Criteria:

* Refusal to participate
* Patients physically or psychologically unable to understand the study and the research protocol
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with glaucoma or ocular hypertonia
Sampling Method: Non-Probability Sample
Enrollment: 1528 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Modelisation of IOP profile | Baseline
  Modelisation of IOP profile of all surgical techniques and additional procedures during the follow-up

SECONDARY OUTCOMES:
Modelisation of IOP profile of Non-perforating deep sclerectomy | Baseline
  Modelisation of IOP profile of Non-perforating deep sclerectomy
Modelisation of IOP profile of Trabeculectomy | Baseline
  Modelisation of IOP profile of Trabeculectomy
Modelisation of IOP profile of Glaucoma drainage device | Baseline
  Modelisation of IOP profile of Glaucoma drainage device
Modelisation of IOP profile of MIGS Istent | Baseline
  Modelisation of IOP profile of MIGS Istent
Modelisation of IOP profile of MIGS XEN | Baseline
  Modelisation of IOP profile of MIGS XEN
Modelisation of IOP profile of High Intensity Focused ultrasound | Baseline
  Modelisation of IOP profile of High Intensity Focused ultrasound
Modelisation of IOP profile of CycloDiode | Baseline
  Modelisation of IOP profile of CycloDiode

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No